CLINICAL TRIAL: NCT05683236
Title: The Clinical Effect Evaluation of Multidisciplinary Collaborative Team Combined With Palliative Care Model in Patients With Terminal Cancer: A Randomised Controlled Study
Brief Title: The Clinical Effect of Palliative Treatment on Patients With Terminal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shijiazhuang People's Hospital (Other)
Responsible Party: Principal Investigator, Yujing Liu, head nurse, Shijiazhuang People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ShijiazhuangPeoplesH
Record Dates: First submitted 2022-12-25; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Multidisciplinary Collaborative; Palliative Care Model; Quality of Life
MeSH Terms: interventions — Patient Comfort

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The patients in the intervention group received multidisciplinary collaborative team care combined with palliative care.
  Interventions: Other: Health education; Other: Comfort care; Other: Pain care; Other: Dietary care; Other: Psychological and social support care
- control group (Active Comparator): The control group was given routine nursing intervention.
  Interventions: Other: routine nursing intervention

INTERVENTIONS:
Other: Health education — Doctors carried out health education for patients to avoid patients giving up their lives, encouraged them to actively cooperate with medical staff, and instructed patients on how to face the disease with a brave and strong attitude and actively fight the disease. Nurses conducted daily psychological counselling for patients, learnt their inner thoughts through communication with patients, and provided timely comfort and encouragement. An attention-shifting method can be used to alleviate the patient's attention to the disease, effectively improving internal depression and avoiding depression. For patients with anxiety and loneliness, family members were instructed to accompany and care.
  Arms: intervention group
Other: Comfort care — Reasonable control of indoor temperature and humidity is necessary to ensure that warm, light conditions permit properly dressed patients to feel warm. Nurses need to ensure that patients are kept clean and tidy in personal hygiene. They would regularly assist patients in turning over while giving patients sufficient respect.
  Arms: intervention group
Other: Pain care — Clinicians should regularly evaluate the patient's physical pain and give reasonable analgesic drugs to patients. Nurses should closely observe the medication response of patients. At the same time, it is necessary to observe and record patients' physical pain daily and take effective pain control measures.
  Arms: intervention group
Other: Dietary care — The clinical nutritionist formulated appropriate nutritional diets according to the nutritional status and personal preferences of patients, provided nutritional support for patients, and followed up with patients once a week after discharge to improve their nutritional status.
  Arms: intervention group
Other: Psychological and social support care — Two nurses with psychological counselling qualifications in the team used the anxiety and depression scale to evaluate the psychological and emotional status of patients and referred to "The Questionnaire Survey on Awareness of Palliative Care" by the Department of Elderly Section of the union medical college hospital. The content mainly included the patient's medical history and general situation, the needs and awareness of patients and their families for palliative care, the choice of patients and their families for the final treatment plan, and the needs of families for grief counselling. Timely professional counselling and intervention were undertaken to alleviate the patient's adverse emotions.
  Arms: intervention group
Other: routine nursing intervention — The control group was given routine nursing intervention, strictly in accordance with a routine treatment process, monitoring the vital signs of patients, giving basic nursing, health education, diet guidance and so on.
  Arms: control group

SUMMARY:
This study proposed a multidisciplinary collaborative team combined with a palliative care model and proposed to establish a team composed of medical staff in various disciplines to make up for the defects of a conventional nursing team. This study applied the multidisciplinary collaboration team combined with a palliative care model to patients with terminal cancer to evaluate its clinical effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients were diagnosed as terminal by imaging, pathology and clinical manifestations
* the expected length of stay was more than seven days
* patients with clear consciousness, good communication and understanding ability
* voluntary participation in this study and signing of informed consent
* the estimated survival period is more than three months

Exclusion Criteria:

* Patients with cognitive impairment and mental illness
* those who were seriously ill and could not cooperate with the completion
* patients with severe communication disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Self-rating Anxiety Scale | Within 8 hours after hospitalization
  This involved 20 items, of which the 5th, 9th, 13th, 17th and 19th items were reverse scoring, and the 1-5 items were positive scoring. The items were scored according to Likert4 grade. The sum of the scores of each item is the total score of the scale. The scores were converted to a standard score: standard score = total anxiety score×1.25. The higher the score, the more severe the anxiety state. A score <50 showed no anxiety, 50-59 showed mild anxiety, 60-69 showed moderate anxiety, and >70 showed severe anxiety
Self-rating Anxiety Scale | through study completion, an average of 1 year
  This involved 20 items, of which the 5th, 9th, 13th, 17th and 19th items were reverse scoring, and the 1-5 items were positive scoring. The items were scored according to Likert4 grade. The sum of the scores of each item is the total score of the scale. The scores were converted to a standard score: standard score = total anxiety score×1.25. The higher the score, the more severe the anxiety state. A score <50 showed no anxiety, 50-59 showed mild anxiety, 60-69 showed moderate anxiety, and >70 showed severe anxiety
Self-rating Depression Scale | Within 8 hours after hospitalization
  There are a total of 20 entries, of which 10 are scored by forward and 10 by reverse. The entries are scored by Likert4 level. The sum of the scores of each item is the total score of the scale. The scores were converted to a standard score: standard score = total anxiety score×1.25. The higher the score, the more serious the depression. A score ≤50 showed no depression, 50-59 showed mild depression, 60-69 showed moderate depression, and >70 showed severe depression
Self-rating Depression Scale | through study completion, an average of 1 year
  There are a total of 20 entries, of which 10 are scored by forward and 10 by reverse. The entries are scored by Likert4 level. The sum of the scores of each item is the total score of the scale. The scores were converted to a standard score: standard score = total anxiety score×1.25. The higher the score, the more serious the depression. A score ≤50 showed no depression, 50-59 showed mild depression, 60-69 showed moderate depression, and >70 showed severe depression
Social Support Rating Scale | Within 8 hours after hospitalization
  The scale was with a total of 10 items, including three dimensions of subjective support, objective support and utilisation of support. The total score of the scale is the sum of the scores of the three dimensions, and the higher the score, the greater the social support. Judgement criteria: A total score of ≤22 indicates a low level, 23-44 indicates a moderate level, and 45-66 indicates a high level, with a domestic norm score of 34.56±3.73
Social Support Rating Scale | through study completion, an average of 1 year
  The scale was with a total of 10 items, including three dimensions of subjective support, objective support and utilisation of support. The total score of the scale is the sum of the scores of the three dimensions, and the higher the score, the greater the social support. Judgement criteria: A total score of ≤22 indicates a low level, 23-44 indicates a moderate level, and 45-66 indicates a high level, with a domestic norm score of 34.56±3.73
Quality of Life Scale | Within 8 hours after hospitalization
  QLQ-C30 consists of one overall QOL scale and five functional scales. The functional scales include physical function, role function, emotional function, cognitive function and social function. Rating criteria: After the scores of each part of the scale are converted to standardised scores, and the score range is 0-100. The higher the score on the scale, the better the overall QOL and functional status
Quality of Life Scale | through study completion, an average of 1 year
  QLQ-C30 consists of one overall QOL scale and five functional scales. The functional scales include physical function, role function, emotional function, cognitive function and social function. Rating criteria: After the scores of each part of the scale are converted to standardised scores, and the score range is 0-100. The higher the score on the scale, the better the overall QOL and functional status

CONTACTS AND LOCATIONS:
Locations (1):
- Shijiazhuang People's Hospital, Shijiazhuang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu YJ, Wu LP, Wang H, Han Q, Wang SN, Zhang J. The clinical effect evaluation of multidisciplinary collaborative team combined with palliative care model in patients with terminal cancer: a randomised controlled study. BMC Palliat Care. 2023 Jun 13;22(1):71. doi: 10.1186/s12904-023-01192-7. PMID 37312118